CLINICAL TRIAL: NCT01549197
Title: End-of-life in French Intensive Care Units: Perception of the Quality of Dying and Experience of Physicians, Nurses and Relatives. Validation of the CAESAR Scale
Brief Title: Quality of Dying in the Intensive Care Unit: Validation of the CAESAR Scale
Acronym: CAESAR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM10104
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Anxiety; Depression; Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU staff and relatives

SUMMARY:
The purpose of the study is to evaluate the quality of the dying process in french ICUs (assessed by the CAESAR scale) and to compare physicians', nurses' and relatives perceptions and experiences, with a one-year follow-up of bereaved relatives.

Our hypothesis is that perception of the quality of dying may impact on relatives' experience of bereavement (anxiety, depression, complicated grief, posttraumatic stress disorder (PTSD)).

DETAILED DESCRIPTION:
Seventy percent of all deaths occur in the hospital environment, and amongst them 20% occur in intensive care units (ICU). In France, no studies have evaluated the quality of the end-of-life process from both the professional and the lay perspective.

The CAESAR scale has been developed from literature reviews and qualitative interviews with relatives, physicians and nurse to assess quality of dying in ICU. Our hypothesis is that perception of the quality of dying may impact on relatives' experience of bereavement (anxiety, depression, complicated grief, PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients Deceased in the ICU after at least 48 hours of ICU stay
* At least one visit of a relative in the ICU

Exclusion Criteria:

* no French-speaking relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians and nurses in charged of ICU deceased patients Bereaved relatives of ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
CAESAR score | Within 3 weeks after patient's death
  Score on the 32-item CAESAR scale assessing quality of end-of-life process

SECONDARY OUTCOMES:
Job strain of the physicians and nurses in charge of the patient | within 3 weeks following patient's death
  Score on the Job strain, a validated scale assessing stress in work environment
Anxiety and depression | 3 months after patient's death
  Anxiety and depression of the relative, assessed by the Hospital Anxiety and Depression Scale (HADS)
Post Traumatic Stress Disorder | 3 months after patient's death
  PTSD of relatives assessed by Inventory of Event Scale revised (IES-R)
Complicated Grief | 6 months after patients' death
  Complicated grief assessed by the Inventory of Complicated Grief (ICG) scale
PTSD | 6 months after patient's death
  PTSD assessed by IES-R
PTSD | 12 months after patient's death
  PTSD assessed by IES-R

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Kentish-Barnes, PhD, Principal Investigator — Reanimation Médicale, Hôpital Saint Louis
Locations (47):
- France (47):
  - Réanimation médicale Centre hospitalier Pays d'Aix, Aix-en-Provence
  - Réanimation Polyvalente Centre Hospitalier Victor Dupouy, Argenteuil
  - Réanimation médicale Hôpital Saint André, Bordeaux
  - Réanimation médicale CHU de la Cavale Blanche, Brest
  - Réanimation Chirurgicale, Caen
  - Réanimation Médicale Hôpital de Caen, Caen
  - Réanimation Médico-Chirugicale CH Chambéry, Chambéry
  - Réanimation CHU ESTAING, Clermont-Ferrand
  - Réanimation polyvalente CH de Dieppe, Dieppe
  - Réanimation polyvalente CH Sud Francilien, Évry
  - Réanimation Polyvalente Centre Hospitalier de Gonesse, Gonesse
  - Réanimation polyvalente Hôpital Les Oudairies, La Roche-sur-Yon
  - Réanimation polyvalente Centre hospitalier de Versailles, Le Chesnay
  - Réanimation médicale Hôpital Calmette, Lille
  - Réanimation polyvalente Hôpital Roger Salengro, Lille
  - Réanimation polyvalente CH Bretagne Sud, Lorient
  - Réanimation médicale Hôpital de La Croix Rousse, Lyon
  - Réanimation Médicale Groupement Hospitalier Edouard Herriot, Lyon
  - Réanimation polyvalente GH Edouard Herriot, Lyon
  - Service de réanimation Institut Paoli Calmettes, Marseille
  - Service d'anesthésie et de réanimation Chu Timone, Marseille
  - Service d'anesthésie et de réanimation Hôpital Nord, Marseille
  - Service de réanimation, détresses respiratoires et infections sévères Hôpital Nord, Marseille
  - Réanimation Centre hospitalier Marc Jacquet, Melun
  - Réanimation Anesthésie CHU Saint Eloi, Montpellier
  - Réanimation Centre Hospitalier Intercommunal André Grégoire, Montreuil
  - Réanimation médicale CHU de Nancy- Hôpital central, Nancy
  - Anesthésie-Réanimation CHU de Nantes- Hôtel Dieu, Nantes
  - réanimation chirurgicale Groupe Hospitalier Universitaire Carémeau, Nîmes
  - Service de réanimation polyvalente CHR - Hôpital de la Source, Orléans
  - Reanimation medicale, Hôpital Saint Louis, Paris
  - Neuro-réanimation chirurgicale Groupe hospitalier Pitié-Salpêtrière, Paris
  - Service de réanimation Hôpital Saint Joseph, Paris
  - Réanimation chirurgicale Hôpital Saint-Louis, Paris
  - Service de réanimation médicale et toxicologique CHU Lariboisière, Paris
  - Réanimation médicale Hôpital Cochin, Paris
  - Réanimation polyvalente au CH d'Annecy, Pringy
  - Réanimation médico-chirurgicale CH de Roanne, Roanne
  - Service de réanimation médicale Hôpital Victor Provo, Roubaix
  - Service de réanimation médicale CHU CH Nicolle, Rouen
  - Service de réanimation polyvalente CH de Saint Lô, Saint-Lô
  - Réanimation polyvalente Centre hospitalier d'Angoulême, Saint-Michel
  - Réanimation Hôpital Font-Pré, Toulon
  - Réanimation médicale Hôpital Chatilliez, Tourcoing
  - Service de réanimation polyvalente CH de Valenciennes, Valenciennes
  - Réanimation Polyvalente CH Bretagne Atlantique, Vannes
  - Service de réanimation médico-chirurgicale Institut Gustave Roussy, Villejuif